CLINICAL TRIAL: NCT05484102
Title: Preventive Effect of Cow's Milk Fermented With Lactobacillus Paracasei CBA L74 on Upper Respiratory Tract and Gastrointestinal Infectious Diseases in Children: a Double-blind, Randomized, Placebo-controlled Trial
Brief Title: Preventive Effect of Cow's Milk Fermented With Lactobacillus Paracasei CBA L74 on Common Infectious Diseases in Children
Acronym: FERCT19
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Bari (Other)
Collaborators: Heinz Italia SpA (Industry)
Responsible Party: Principal Investigator, Ruggiero Francavilla, Professor, University of Bari
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: FERCT19
Record Dates: First submitted 2020-09-27; First posted 2022-08-02 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Upper Respiratory Tract Infections; Gastrointestinal Infection; Children, Only
Keywords: Lactobacillus paracasei CBA L74; fermented milk
MeSH Terms: conditions — Respiratory Tract Infections

STUDY DESIGN:
Intervention Model Description: double blind randomized placebo controlled clinical trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Enrolled children will be randomly assigned, with the use of a computer-generated randomization list to receive milk fermented with Lactobacillus paracasei CBA L74 or placebo
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- lactobacillus paracasei CBA L74 (Experimental): 100 enrolled children will receive milk fermented with lactobacillus paracasei CBA L74 daily for 3 months.
  Interventions: Dietary Supplement: milk fermented with lactobacillus paracasei CBA L74
- placebo (Placebo Comparator): 100 enrolled children will receive placebo milk formula containing maltodextrins daily for 3 months.
  Interventions: Dietary Supplement: placebo milk formula

INTERVENTIONS:
Dietary Supplement: milk fermented with lactobacillus paracasei CBA L74 — milk fermented with lactobacillus paracasei CBA L74 will be administered daily for 3 months to 100 children. Participants were supplied with the milk product in powder form, by Heinz Italia SpA, Segrate, Italy. The study products were provided in tins containing 400 g of powder, and the packaging was similar and the tins were stored at room temperature in a dry environment. The family pediatricians instructed parents about the daily amount of the assigned study product and the method of preparation. All subjects received 7 g/day of study products diluted in a maximum of 150 mL of cow's milk or water. After dilution, the look and the taste were the same for all of the study products.
  Arms: lactobacillus paracasei CBA L74
Dietary Supplement: placebo milk formula — placebo milk formula containing maltodextrins will be administered daily for 3 months to 100 children. The study products were provided in tins containing 400 g of powder, and the packaging was similar and the tins were stored at room temperature in a dry environment. The family pediatricians instructed parents about the daily amount of the assigned study product and the method of preparation. All subjects received 7 g/day of study products diluted in a maximum of 150 mL of cow's milk or water. After dilution, the look and the taste were the same for all of the study products.
  Arms: placebo

SUMMARY:
this is a double-blind randomized placebo controlled clinical trial. 200 healthy children aged 12-48 months, attending day care or preschool for at least 5 days a week, regularly checked by the family pediatrician (FP) involved in the trial, were considered for the study and consecutively contacted during scheduled medical examinations at the FPs office. study plan is 3-month treatment period. The clinical evaluation will be carried out at enrollment, at 30, 60 and 90 days from the beginning of the treatment by the pediatrician. fecal and nasal mucus samples for immunological and microbiological analysis will be collected before the treatment and at 90 days (end of treatment).

DETAILED DESCRIPTION:
Subjects were supplemented daily for 3 months with cow's skim milk fermented with L. paracasei CBA L74 (group A) or placebo (group B).Enrolled children will be randomly assigned, with the use of a computer-generated randomization list to receive either milk fermented with Lactobacillus paracasei CBA L74 or placebo once. Placebo and fermented milk had the same shape, the placebo's taste, dimension, indication, and appearance. At enrollment the family pediatricians consulted the clinical records of each child for previous diseases and pharmacological treatments. At the baseline, after obtaining informed consent from the parents/tutors of each child, the health status of all the study subjects was carefully assessed, and the presence of infectious diseases or other disease was ruled out by means of a complete physical examination, including vital signs (body temperature, pulse rate, respiration rate, blood pressure); neurological status; body growth status; nutritional status; hydration; skin evaluation; otoscopy; evaluation of oral cavity; respiratory/abdomen/lymphonode examination; and genital examination.

A diary will be given to the parents; on a daily basis, patients will monitor and record the frequency/severity of symptoms, episodes of respiratory and/or gastrointestinal infection and their duration and school absence on the diary.

Fecal Analysis: three fecal samples for microbiological and immunological analysis will be collected before treatment and at 90 days (end of treatment). Nasal mucus samples for immunological analysis will be collected before the treatment and at 90 days (end of the treatment).

The study was approved by the Ethics Committee of the Universities of Bari.

ELIGIBILITY:
Inclusion Criteria:

* Healthy children aged 12-48 months
* attending day care or preschool for at least 5 days a week

Exclusion Criteria:

The exclusion criteria were:

* age <12 months or >48 months
* concomitant chronic infections, chronic systemic diseases, chronic inflammatory bowel diseases, autoimmune diseases, immunodeficiency, malignancy, metabolic diseases
* chronic respiratory tract diseases including respiratory allergies and cystic fibrosis
* malformations of gastrointestinal or urinary or respiratory tract
* history of respiratory or gastrointestinal or urinary tract surgery
* congenital cardiac defects
* functional bowel disorders
* suspected or challenge-proved food allergy, food intolerances
* severe malnutrition (z-score for weight-for-height <3 standard deviation scores)
* use of antibiotics or pre/pro/synbiotics or immune stimulating products in the 2 weeks before the enrolment
* Siblings of subjects enrolled in the study were not allowed to participate to the trial.

Ages: 12 Months to 48 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 200 (Actual)
Dates: Start 2022-09-15 (Actual); Primary Completion 2024-01-10 (Actual); Study Completion 2024-01-11 (Actual)

PRIMARY OUTCOMES:
preventive effect of cow's milk fermented with Lactobacillus paracasei CBA L74 on common infectious disease | 3 months
  the rate of children experiencing at least one episode of common infectious disease

SECONDARY OUTCOMES:
Total number of common infectious disease | 3 months
  evaluate the total number of common infectious disease
use of medications | 3 months
  use of medications (antibiotics, antipyretics, steroids)
emergency department medical examinations and hospitalizations | 3 months
  access to emergency department medical examinations and hospitalizations
days of work lost by the parents | 3 months
  evaluation of days of work lost by the parents
days of school lost by the children | 3 months
  evaluation of days of school lost by the children

CONTACTS AND LOCATIONS:
Overall Officials: ruggiero francavilla, Principal Investigator — University of Bari
Locations (1):
- Clinica Pediatrica, Bari, Apulia, Italy

IPD SHARING:
Plan to Share IPD: No
The investigators were blinded to the treatment at all times (i.e., allocation, intervention, laboratory analysis and statistical analysis). The study subjects were allocated to two groups (group A or group B) according to a computer-generated randomization list. The pediatricians, parents, and the children were blinded to the allocated treatment. Subjects were supplemented daily for 3 months with cow's skim milk fermented with L. paracasei CBA L74 (group A) or placebo (group B).

REFERENCES:
- [Result] Maldonado J, Canabate F, Sempere L, Vela F, Sanchez AR, Narbona E, Lopez-Huertas E, Geerlings A, Valero AD, Olivares M, Lara-Villoslada F. Human milk probiotic Lactobacillus fermentum CECT5716 reduces the incidence of gastrointestinal and upper respiratory tract infections in infants. J Pediatr Gastroenterol Nutr. 2012 Jan;54(1):55-61. doi: 10.1097/MPG.0b013e3182333f18. PMID 21873895
- [Result] Tamang JP, Shin DH, Jung SJ, Chae SW. Functional Properties of Microorganisms in Fermented Foods. Front Microbiol. 2016 Apr 26;7:578. doi: 10.3389/fmicb.2016.00578. eCollection 2016. PMID 27199913
- [Result] Tamang JP, Watanabe K, Holzapfel WH. Review: Diversity of Microorganisms in Global Fermented Foods and Beverages. Front Microbiol. 2016 Mar 24;7:377. doi: 10.3389/fmicb.2016.00377. eCollection 2016. PMID 27047484
- [Result] Hill C, Guarner F, Reid G, Gibson GR, Merenstein DJ, Pot B, Morelli L, Canani RB, Flint HJ, Salminen S, Calder PC, Sanders ME. Expert consensus document. The International Scientific Association for Probiotics and Prebiotics consensus statement on the scope and appropriate use of the term probiotic. Nat Rev Gastroenterol Hepatol. 2014 Aug;11(8):506-14. doi: 10.1038/nrgastro.2014.66. Epub 2014 Jun 10. PMID 24912386
- [Result] Perna A, Intaglietta I, Simonetti A, Gambacorta E. Effect of genetic type and casein haplotype on antioxidant activity of yogurts during storage. J Dairy Sci. 2013 Jun;96(6):3435-41. doi: 10.3168/jds.2012-5859. Epub 2013 Mar 30. PMID 23548278
- [Result] Merenstein D, Murphy M, Fokar A, Hernandez RK, Park H, Nsouli H, Sanders ME, Davis BA, Niborski V, Tondu F, Shara NM. Use of a fermented dairy probiotic drink containing Lactobacillus casei (DN-114 001) to decrease the rate of illness in kids: the DRINK study. A patient-oriented, double-blind, cluster-randomized, placebo-controlled, clinical trial. Eur J Clin Nutr. 2010 Jul;64(7):669-77. doi: 10.1038/ejcn.2010.65. Epub 2010 May 19. PMID 20485304
- [Result] Brunser O, Araya M, Espinoza J, Guesry PR, Secretin MC, Pacheco I. Effect of an acidified milk on diarrhoea and the carrier state in infants of low socio-economic stratum. Acta Paediatr Scand. 1989 Mar;78(2):259-64. doi: 10.1111/j.1651-2227.1989.tb11066.x. PMID 2929349
- [Result] Campeotto F, Suau A, Kapel N, Magne F, Viallon V, Ferraris L, Waligora-Dupriet AJ, Soulaines P, Leroux B, Kalach N, Dupont C, Butel MJ. A fermented formula in pre-term infants: clinical tolerance, gut microbiota, down-regulation of faecal calprotectin and up-regulation of faecal secretory IgA. Br J Nutr. 2011 Jun 28;105(12):1843-51. doi: 10.1017/S0007114510005702. Epub 2011 Mar 22. PMID 21426607
- [Result] Nagata S, Asahara T, Ohta T, Yamada T, Kondo S, Bian L, Wang C, Yamashiro Y, Nomoto K. Effect of the continuous intake of probiotic-fermented milk containing Lactobacillus casei strain Shirota on fever in a mass outbreak of norovirus gastroenteritis and the faecal microflora in a health service facility for the aged. Br J Nutr. 2011 Aug;106(4):549-56. doi: 10.1017/S000711451100064X. Epub 2011 Apr 27. PMID 21521545
- [Result] Nocerino R, Paparo L, Terrin G, Pezzella V, Amoroso A, Cosenza L, Cecere G, De Marco G, Micillo M, Albano F, Nugnes R, Ferri P, Ciccarelli G, Giaccio G, Spadaro R, Maddalena Y, Berni Canani F, Berni Canani R. Cow's milk and rice fermented with Lactobacillus paracasei CBA L74 prevent infectious diseases in children: A randomized controlled trial. Clin Nutr. 2017 Feb;36(1):118-125. doi: 10.1016/j.clnu.2015.12.004. Epub 2015 Dec 17. PMID 26732025